CLINICAL TRIAL: NCT02368262
Title: Prevalence of Incontinence and Risk Factors in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/766.2
Record Dates: First submitted 2015-02-13; First posted 2015-02-23 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Urinary Incontinence
Keywords: Cerebral Palsy; Risk factors; Child; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence; Cerebral Palsy | interventions — Surveys and Questionnaires; Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- CP- incontinent: Children with CP and daytime incontinence. Evaluation consisted of a questionnaire and micturition and drinking diaries, uroflowmetry, pelvic floor EMG and bladderscan.
  Interventions: Other: Questionnaire and micturition and drinking diaries; Procedure: Uroflowmetry, pelvic floor EMG and bladderscan
- CP- continent: Children with CP without daytime incontinence. Evaluation consisted of a questionnaire and micturition and drinking diaries, uroflowmetry, pelvic floor EMG and bladderscan.
  Interventions: Other: Questionnaire and micturition and drinking diaries; Procedure: Uroflowmetry, pelvic floor EMG and bladderscan
- NoDev - incontinent: Children with normal development with daytime incontinence. Evaluation consisted of a questionnaire and micturition and drinking diaries, uroflowmetry, pelvic floor EMG and bladderscan.
  Interventions: Other: Questionnaire and micturition and drinking diaries; Procedure: Uroflowmetry, pelvic floor EMG and bladderscan
- NoDev - continent: Children with normal development without daytime incontinence. Evaluation consisted of a questionnaire and micturition and drinking diaries, uroflowmetry, pelvic floor EMG and bladderscan.
  Interventions: Other: Questionnaire and micturition and drinking diaries; Procedure: Uroflowmetry, pelvic floor EMG and bladderscan

INTERVENTIONS:
Other: Questionnaire and micturition and drinking diaries — Questionnaire: ICCS parental questionnaire + extended history taking document, ROME III criteria, demographic information and/or PIN-Q.
  Diaries: 24-hour voiding chart
Procedure: Uroflowmetry, pelvic floor EMG and bladderscan — Voiding variables, pelvic floor activity during micturition and postmictional residue.

SUMMARY:
This study evaluates (risk)factors influencing (in)continence in children with and without a brain injury.

DETAILED DESCRIPTION:
Children with cerebral palsy (CP) (Rosenbaum, 2007) gain bladder and bowel control at older age compared to typical developing children (Ozturk, 2006). The incidence of urinary incontinence during day and night, fecal incontinence and constipation is higher in this population.

Incontinence in children is often treated with urotherapy. This is a nonsurgical, nonpharmacological treatment for lower urinary tract dysfunctions. Standard urotherapy is noninterventional and it includes giving information, instructions, advice regarding life-style, fluid intake and bladder diaries. Additionally specific interventions can be used, such as: various forms of pelvic floor training, behavioral modification, biofeedback, electrical stimulation and catheterization (Neveus, 2006). Recent research has proven urotherapy to be successful for the treatment of children with daytime incontinence (Mulders, 2010).

Despite the high prevalence of incontinence in children with CP the possible treatment strategies in this population are poorly investigated. Far too often, urinary incontinence in children with CP is considered a normal, unavoidable and even a minor problem.

Aim: Analyze (risk) factors influencing (in)continence in children with and without CP.

Possible parameters will be registered through questioning, measurement (uroflow combined with pelvic floor EMG and postmictional residue) and retrospective analysis of the patient files. Parameters will be compared between continent and incontinent children with and without CP. This comparison evaluates whether the same therapeutic strategies can be applied in incontinent children with and without CP.

ELIGIBILITY:
Inclusion Criteria:

* Daytime urinary incontinence with or without enuresis and/or fecal incontinence (Groups with incontinence)
* No urinary or fecal incontinence (Groups without incontinence)
* Cerebral palsy (Groups with children with CP)
* Normal development (Groups with children without CP)

Exclusion Criteria:

* Isolated urinary tract infections
* Isolated enuresis
* Isolated dysfunctional voiding
* Isolated fecal incontinence
* Anatomical abnormalities
* History of genitourinary or renal surgery
* Medication for incontinence during the last 3 months
* Pelvic reeducation during the last 6 months
* Other neurologic problems influencing continence

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with CP: Cerebral palsy Reference Centre (Ghent university hospital) Incontinent children with normal development: Urology department (Ghent university hospital) continent children with normal development: community sample
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Risk factors | Cross-sectional
  Identification of predictive factors for incontinence in children with and without CP.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Van Laecke, PhD MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital, Ghent, Ghent, Belgium